CLINICAL TRIAL: NCT00352781
Title: The STOP (Stop Smoking Therapy for Ontario Patients) Study: The Effectiveness of Nicotine Replacement Therapy in Ontario Smokers PHASE II
Brief Title: Stop Smoking Therapy for Ontario Patients
Acronym: STOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government); Pfizer (Industry)
Responsible Party: Principal Investigator, Dr. Peter Selby, Clinical Director, Addictions Program, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 064/2006
Record Dates: First submitted 2006-07-13; First posted 2006-07-17 (Estimated); Results first posted 2012-04-17 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Smoking
Keywords: nicotine replacement therapy; smoking cessation
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Nicotine Replacement Therapy; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nicotine Replacement + Behaviour Therapy (Experimental): Nicotine Replacement Therapy as per monograph & behavioural intervention
  Interventions: Drug: nicotine replacement therapy; Behavioral: behavioural intervention

INTERVENTIONS:
Drug: nicotine replacement therapy — nicotine transdermal patches as per product monograph
  Other Names: Nicoderm
Behavioral: behavioural intervention — Smoking cessation counselling and relapse prevention

SUMMARY:
Approximately 2 million Ontarians are current smokers. While smoking rates have declined over the past 25 years, these rates have remained constant since 2002. The rate of smoking cessation in Ontario has not kept up with the rest of Canada. A new strategy is necessary to increase the number of smokers making quit attempts and to increase the odds of quitting over the long term.

The overall goal of the Stop Smoking Therapy for Ontario Patients (STOP) Study is to evaluate the methods and effectiveness of providing nicotine replacement therapy (NRT) to Ontario smokers. The study will develop an evidence-based protocol for providing NRT, provide faculty development on combining pharmacotherapy with behavioural interventions and will provide an evaluation framework to inform future coverage models.

The goal for this phase of the STOP study is to provide faculty development on combining pharmacotherapy with behavioural interventions. This will be achieved by partnering with Public Health Units across Ontario who have established smoking cessation clinics but do not have the finances in place to offer NRT to their clients at a subsidized rate or free of charge. Cost has been shown to be a significant barrier to the access and use of NRT in individuals trying to quit smoking. However, combining pharmacotherapy with behavioural interventions may be more effective than either alone. Therefore, we hypothesize that providing NRT free of charge to clients enrolled in a smoking cessation clinic will be more effective for smoking cessation than behavioural interventions alone.

DETAILED DESCRIPTION:
According to the US Surgeon General's Report (1988), there are immediate, intermediate and long-term benefits to health from quitting smoking. For example, there is a 50% reduction in coronary heart disease risk in 12 months and the risk of a stroke is reduced to that of a nonsmoker 5-15 years after quitting. (US Surgeon General's Report, 1990, p.vi).

In a systematic assessment of the value of clinical preventive services recommended by the US Preventive Services Task Force, smoking cessation treatment for adults was one of the highest-ranked services in terms of its cost effectiveness and its potential to reduce the burden of disease. Most smoking cessation interventions cost less per year of life saved than most widely accepted medical practices. For example, cost-effectiveness analysis of the implementation of the Agency for Healthcare Research and Quality (AHRQ) guidelines show costs of $4,113 per life-year saved, in 2001 prices compared to annual mammography for women aged 40 to 49 years, which costs $71,751 in 2001 prices, and hypertension screening for men aged 40 years, which costs $27,117 in 2001 prices. Therefore, smoking cessation services have been referred to as the "gold standard" for comparing the cost effectiveness of other healthcare interventions. Although some studies have shown high costs from increased healthcare utilization in the first year after quitting smoking due to illness (Martinson, 2003), most studies demonstrate that smokers who quit eventually have significantly lower healthcare utilization than continuing smokers (Fishman, 2003; Warner, 2003) Thus, for healthcare organizations such as the Ontario Health Insurance Plan, implementing smoking cessation services will likely result in a relatively quick return on investment.

Both the intensity and duration of behavioural interventions are associated with sustained remission in smoking. The addition of pharmacotherapy doubles the odds of quitting successfully. However, many smokers face barriers in accessing pharmacotherapy. The provision of free pharmacotherapy has the potential to help a substantial number of smokers to quit. A study by Curry et al, 1998, evaluated smokers who were willing to sign up for a cessation-support program under various degrees of coverage for either the program or nicotine replacement therapy (NRT). 10% of Smokers with full coverage were likely to attempt to quit as opposed to 2.5% with partial coverage. Therefore, the United States Health & Human Services guidelines call for the coverage of these medications.

Research has shown that coverage for tobacco dependence treatments can enhance not only the rate of quit attempts but also long-term abstinence for smokers (Levy & Friend, 2002; Schauffler, McMenamin, Olson, Boyce-Smith, Rideout, & Kamil, 2001). On average, the odds ratio of quitting at one year was 1.6 for those given free NRT. Therefore, some insurers, both public and private, reimburse patients for stop smoking medications. However, a study by Boyle et al 2002, found that simply including the medication in an insurance plan did not increase quit rates or utilization of medications. Adequate precautions must be taken to ensure that free pharmacotherapy is distributed in conjunction with behavioural interventions to be successful and to be used by those smokers most likely to benefit from pharmacotherapy.

Pharmacotherapy can be very expensive if provided to all smokers. However, not all smokers want to quit or require medications to quit (McDonald, 2003). Most smokers use about 2-3 weeks of pharmacotherapy when not combined with behavioural interventions (Pierce, 2002). About 0.05% of smokers looking to quit will seek specialized care. Moreover, if we assume that 70% of current tobacco users (Approximately 1.6 million) in Ontario will try to quit in a given year and that 10% ( i.e. 169,000) of these individuals would qualify for and seek reimbursement for 10 weeks of therapy at $30/week, then the total estimated cost will be about $50 million! This is clearly not fundable and therefore a comprehensive strategy combined with some rational use of pharmacotherapy is necessary.

Hypotheses:

1. The provision of free NRT will increase quit attempts in Ontario smokers
2. The provision of free NRT will increase long-term quit rates (>/= 6 months) in Ontario smokers.
3. Smokers who quit smoking using NRT will have reduced health care costs after the first year of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be current residents of Ontario.
* Older than or equal to 18 years of age.
* Current daily smokers who smoke 10 or more cigarettes per day for at least 3 months.
* Has smoked more than 100 cigarettes in their lifetime.

Exclusion Criteria:

* Varenicline treatment, current.
* Intolerant to nicotine replacement therapy (NRT)
* Have a medical condition that would make participation medically hazardous as determined by the list of contraindications for NRT outlined in the Compendium of Pharmaceuticals and Specialties (CPS) and the NRT package insert, including a heart attack in the past two (2) weeks, life-threatening arrhythmias, severe or worsening angina pectoris, recent cerebro-vascular incident (past two (2) weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1767 (Actual)
Dates: Start 2006-07; Primary Completion 2009-01 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Selby, MD, MHSc, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.net/research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by their local public health unit.
Groups:
- Nicotine Replacement Therapy + Counseling: Up to 10 weeks of open-label nicotine replacement therapy (as per product monograph) + counseling
Period: Overall Study
Arm/Group | Nicotine Replacement Therapy + Counseling
Started | 1767
Completed | 884
Not Completed | 883

BASELINE CHARACTERISTICS:
Groups:
- Nicotine Replacement Therapy (NRT): Open-label Nicotine Replacement Therapy + counseling
Arm/Group | Nicotine Replacement Therapy (NRT)
Number analyzed (Participants) | 1767
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 1654
  >=65 years | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 997
  Male | 770
Region of Enrollment [Number; unit: participants]
  Canada | 1767

OUTCOME MEASURES:

1. Primary Outcome: Smoking Cessation
Description: 7-day point prevalence of abstinence
Time Frame: 6 months after end of treatment
Population: Number of participants that completed the 6m follow-up (i.e. per protocol)
Measure: Number; unit: percentage of participants abstinent
Groups:
- Nicotine Replacement Therapy: Open-label nicotine replacement therapy (as per product monograph) plus counseling
Arm/Group | Nicotine Replacement Therapy
Number analyzed (Participants) | 395
percentage of participants abstinent | 29

2. Secondary Outcome: Smoking Cessation
Description: 7-day point prevalence of abstinence
Time Frame: 12 months after end of treatment
Population: Number of participants who completed the 12m follow-up
Measure: Number; unit: percentage of participants abstinent
Arm/Group | Nicotine Replacement Therapy
Number analyzed (Participants) | 442
percentage of participants abstinent | 26

ADVERSE EVENTS:
Groups:
- Nicotine Replacement Therapy + Counseling: Up to 10 weeks of open-label nicotine replacement therapy + counseling
Arm/Group | Nicotine Replacement Therapy + Counseling
Serious Adverse Events (participants affected / at risk) | 2/1767
Other Adverse Events (participants affected / at risk) | 0/1767
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Replacement Therapy + Counseling (N=1767)
myocardial infarction (Cardiac disorders) | 1 (1) — Not determined to be related to study medication. Patient used the nicotine patch for one day. Discontinued use after experiencing shortness of breath. Three days after discontinuing patch had an MI.
seizure (Nervous system disorders) | 1 (1) — Unrelated to study medication (nicotine patch). Patient was witnessed having a "seizure" (full body shaking) by a friend. Patient refused to go to the hospital. When followed-up by physician, was not advised to discontinue nicotine patch.

LIMITATIONS AND CAVEATS:
Many participants could not be reached 6 and 12 months after treatment to complete the follow-up questionnaires. Data pertaining to smoker and provider satisfaction and healthcare utilization were not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes